CLINICAL TRIAL: NCT06731413
Title: Phase 2 Study to Evaluate Reduced Dose Chemotherapy in Combination With Anti-PD-1 Therapy as First Line Treatment in Vulnerable or Older Adults (Vulnerable or Age ≥70) With Advanced PD-L1 TPS <50% Non-small Cell Lung Cancer
Brief Title: Reduced CT + Anti-PD-1 as First Line Tx in Vulnerable Older Adults w/Adv <50% PD-L1 Non-Small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-24-21788
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Lung Cancer; NSCLC; Advanced Non-Small Cell Lung Cancer; Metastatic Non Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Reduced Dose Combination Therapy (Experimental): Squamous cell histology:
  1. Carboplatin AUC 3 every 21 days IV for 4 cycles
  2. Paclitaxel 135 mg/m2 every 21 IV days for 4 cycles
  3. Pembrolizumab 200 mg every 21 days IV until disease progression or unacceptable toxicity up to 35 cycles
  Non-squamous histology:
  1. Carboplatin AUC 3 every 21 days IV for 4 cycles
  2. Pemetrexed 375 mg/m2 every 21 IV days for 4 cycles
  3. Pembrolizumab 200 mg every 21 days IV until disease progression or unacceptable toxicity up to 35 cycles
  Interventions: Drug: Reduced Dose of Chemotherapy and Immunotherapy

INTERVENTIONS:
Drug: Reduced Dose of Chemotherapy and Immunotherapy — Eligible participants with recurrent or metastatic squamous cell carcinoma will receive 4 cycles of carboplatin area under the curve (AUC) 3 IV every 21 days and paclitaxel 135 mg/m2 intravenous (IV) every 21 days. Participants with non-squamous histology will receive carboplatin AUC 3 IV every 21 days and pemetrexed 375 mg/m2 IV every 21 days (collectively, induction chemotherapy). Both groups will receive pembrolizumab 200 mg IV every 21 days for a total of up to 35 cycles (Cycles ≥5 are collectively the maintenance portion of treatment) or until disease progression or unacceptable toxicity.

SUMMARY:
Evaluate frequency of adverse events that lead to chemotherapy discontinuation in vulnerable older adults with recurrent/metastatic PD-L1 TPS<50% NSCLC patients who receive reduced dose chemotherapy in combination with immunotherapy.

DETAILED DESCRIPTION:
This is a single institution, single arm, open label phase 2 study in vulnerable or older adults (Age ≥70) with recurrent or metastatic, histologically confirmed squamous cell carcinoma or non-squamous cell carcinoma of lung without driver mutation and PD-L1 TPS < 50% to evaluate safety and tolerability of reduced dose of chemotherapy and immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC) (either squamous or non- squamous)
* Stage IV disease OR have recurrent disease and not be candidates for curative treatment such as combined chemo-radiation
* No previous line of treatment in the recurrent or metastatic setting. Neoadjuvant or adjuvant treatment more than 6 months before enrollment is acceptable.
* Age 70 or meeting frailty definition or above at the date of signing informed consent
* Absence of driver mutations that have first line Food and Drug Administration (FDA) approved targeted therapy
* PD-L1 tumor proportion score (TPS) of less than 50%
* Eastern Cooperative Oncology Group (ECOG) PS of 0-3
* Have measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment
* Absolute neutrophil count (ANC) ≥ 1,000/μL
* Platelets ≥ 75,000/μL
* Hemoglobin (Hgb) ≥ 8.0 g/dL (transfusion permitted)
* Total bilirubin ≤ 2 x institutional upper limit of normal (ULN)
* Aspartate amino transferase (AST)serum glutamic-oxaloacetic transaminase (SGOT) /alanine aminotransferase (ALT)serum glutamic-pyruvic transaminase (SGPT) ≤ 5.0 × institutional ULN
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants with life expectancy of less than 3 months at the time of enrollment
* Has active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, or immunosuppressive drugs)
* Diagnosis of interstitial lung disease
* Creatinine clearance of <30 mL/min
* Symptomatic, untreated central nervous system (CNS) disease or leptomeningeal disease. Patients with asymptomatic or treated CNS disease are eligible
* Required ongoing use of immunosuppressive medication, including steroids, with the following allowable exceptions:

  * Doses less than or equal to the equivalent of prednisone 10 mg daily
  * Short courses of steroids that are discontinued prior to enrollment
  * Inhaled, intranasal and/or topical steroids
  * Dexamethasone taper for treating vasogenic edema associated with CNS disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2033-07-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of chemotherapy discontinuation due to treatment-related adverse events | Through completion of protocol therapy, up to 2 years
  Evaluate treatment tolerability i by the number of participants that discontinue chemotherapy treatment due to treatment-related adverse events.

SECONDARY OUTCOMES:
Response (complete response and partial response) per Response Evaluation Criteria in Solid Tumors | Up to 5 years
  Evaluate overall response defined by complete and partial response in vulnerable or older adults with recurrent/metastatic PD-L1 TPS <50% NSCLC patients who receive reduced dose chemotherapy in combination with immunotherapy per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Overall incidence and severity of all adverse events assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | Time of patient consent and throughout the duration of the study, including during the treatment period and for 30 days following the final dose of the study medication, up to 2 years and 1 month
  The total number of AE's recorded for the protocol.
Overall survival defined as the time from the date of first study treatment until the date of death. Overall survival (OS) will be censored on the last date a participant was known to be alive | Up to 5 years
  Overall survival of participants measured in days.
Progression-free survival (PFS) measured from the date of first study treatment until the date of documented disease progression | Up to 5 years
  Evaluate progression-free survival of participants in days utilizing RECIST 1.1 criteria or death from any cause, whichever occurs first.
Cancer related symptoms and quality of life | Baseline, Cycle 3 Day 1, Cycle 5 Day 1 Cycle 9 Day 1, EOT Visit (up to 2 years)
  Evaluate impact of the reduced dose combination therapy on quality of life as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC-QLQ C30). The EORTC QLG Core Questionnaire (EORTC QLQ-C30) is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients.The functioning and the global QoL scales, a higher score indicates better health. Response options are on a 4-point Likert-type scale (not at all; a little; quite a bit; very much) and a 7-point Likert scale for global HRQoL ranging from 'Very poor' to 'Excellent'. The QLQ-C30 summary score is calculated as the mean of the combined 13 QLQ-C30 scale and item scores with a higher score indicating a better HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Berkman, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Currently there are no plans to share IPD with other researchers.